CLINICAL TRIAL: NCT02885922
Title: The Effects of add-on Anti-diabetic Drugs on Inflammation and Energy Homeostasis in Type 2 Diabetic Patients
Brief Title: The Effects of add-on Anti-diabetic Drugs in Type 2 Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CG16183A
Record Dates: First submitted 2016-08-26; First posted 2016-09-01 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The genetic studies will be applied for efficacy and adverse effect of anti-diabetic drugs.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: anti-diabetic drug — Add-on anti-diabetic drug in type 2 diabetic patients
  Other Names: Glucose lowering

SUMMARY:
Recently, there are some new classes of anti-diabetic drugs availible in Taiwan. In this study, we will observe the change in inflammation and energy homeostasis in type 2 diabetic outpatient, who receiving a new anti-diabetic drugs.

DETAILED DESCRIPTION:
Recently, there are some new classes of anti-diabetic drugs availible in Taiwan. However, the effects of these anti-diabetic drugs should be further evaluated. Specially, the effects on inflammation and energy homeostasis are still not well assessed. In this study, we will observe the change in inflammation and energy homeostasis in type 2 diabetic outpatient, who receiving a new anti-diabetic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic outpatient

Exclusion Criteria:

* Refusal of anti-diabetic drugs
* Preganacy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic patients in Taichung Veterans General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2016-09; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 3 months

SECONDARY OUTCOMES:
Brain-Derived Neurotrophic Factor (BDNF) | 3 months
  energy homeostasis
Body-composition | 3 months
  energy homeostasis
Fasting glucose | 3 months
Hypoglycemia | 3 months
Vascular Cell Adhesion Molecule 1 (VCAM-1) | 3 months
  inflammation
Ankle-Brachial Index (ABI) | 12 months
  peripheral artery disease
Orexin-A | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: I-Te Lee, MD,PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- outpatient clinic of the Division of Endocrinology and Metabolism in Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available